CLINICAL TRIAL: NCT02096198
Title: 36mm CERAMAX® Ceramic Hip System PMA PAS: Long-Term Follow-up of Previously Enrolled Investigational Device Exemption (IDE) Study Subjects
Brief Title: Ceramic On Ceramic (COC) 36mm PAS IDE Rollover Subjects; Ceramic Acetabular Bearing With Ceramic Femoral Head in Total Hip Replacement
Acronym: COC36mmPAS
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 11013
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Avascular Necrosis; Post-Traumatic Osteoarthritis of Hip
Keywords: Total Hip Replacement; Total Hip Arthroplasty; Hip Joint Replacement; Hip Prosthesis Replacement
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Other CERAMAX COC 36mm Acetabular Cup: The CERAMAX COC 36mm ceramic acetabular bearing insert component is manufactured from high purity, dense alumina matrix composite ceramic. The insert is available in several inner diameter sizes, including 36mm; only 36mm inserts will be utilized in this PAS. The inserts secure to DePuy's Pinnacle acetabular shells by means of an interlocking mechanical taper.

SUMMARY:
This study is intended to gather medium (5- to 7-years) and long-term (minimum 8- to 10-years) information regarding the performance and safety of the commercially available 36mm CERAMAX® Ceramic on Ceramic (COC) Total Hip System from a cohort of study subjects that were previously enrolled in the IDE study. (COC = 36mm ceramic acetabular bearing insert component that articulates with a ceramic femoral head in the COC total hip replacement system)

DETAILED DESCRIPTION:
Up to five (5) sites will participate. These sites participated in the IDE study and will continue subject follow-up.

Subjects from the original IDE study (COC 36mm investigational subjects only) will be seen for a clinic visit at the time of consent (First visit at approximately 5 to 7 years post-op or 1825- 2919 days), and at minimum 8 years (2920-3649 days) , and minimum 10 years (3650-4015 days). Harris Hip evaluation, radiographic evaluation, subject hip-outcomes, and adverse event information will be collected at each visit.

If a subject is not willing or able to return for a clinical and radiographic follow-up for either the minimum 8 year evaluation or the minimum 10 year evaluation, then a telephone interview may be utilized for the purpose of determining device survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously enrolled in the COC 36 IDE study;
* Individuals who are willing and able to provide informed patient consent for participation in the study;
* Individuals who are willing and able to return for follow-up as specified by the study protocol; and
* Individuals who are willing and able to complete the Subject Hip Outcomes questionnaire as specified by the study protocol.

Exclusion Criteria:

* In the opinion of the Investigator, the individual does not qualify if there are any concerns with the ability to follow the protocol specified evaluations.
* Any component of the primary total hip was previously revised.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from the original IDE study who have already been implanted with a Ceramax 36mm ceramic-on-ceramic system and who have given their consent for this study
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Device survivorship at 10-years post-operatively | 10-years post-operatively
  Device survivorship will be estimated with a Kaplan-Meier survivorship analysis at 10-years post-operatively.

SECONDARY OUTCOMES:
Harris Hip scores | Harris Hip score means and Harris Hip sub-score means will be estimated at the First visit at 5-7 years (1825- 2919 days); Minimum 8-years (2920-3649 days); Minimum 10-years (3650-4015days)
  The Harris Hip score consists of five sub-scales: Pain, Function, Activities Deformity and Range of motion. The instrument is designed for completion by a clinician.
Subject Hip Outcomes | Subject Hip Outcomes will be estimated at the First visit at 5-7 years (1825- 2919 days); Minimum 8-years (2920-3649 days); Minimum 10-years (3650-4015days)
  Subject Hip Outcomes is a standardized instrument for use as a measure of health outcome that is designed for completion by the study subject. This hips outcomes self-assessment includes five (5) questions about subject satisfaction and hip function. The 5 questions relate to study subject function, pain, need for pain meds, satisfaction and their status (i.e., better, same or worse).
  The percent of subjects who answer 'Yes' or 'Better' on each respective question will be reported.
Radiographic | At first visit (5-7 years), at Minimum 8-years (2920-3649 days); Minimum 10-years (3650-4015 days)
  At 5 to 7 years, at Minimum 8-years and at minimum 10-years, secondary radiographic outcome measures will include high quality antero-posterior and lateral radiographs of the operative hip, which will be obtained during the same postoperative follow-up intervals as for the clinical evaluations. At the first "enrollment" visit (5-7 years), an additional Cross-Table Lateral films will be collected to permit assessment of cup positioning.
  Radiographic views will include:
  * AP Pelvis
  * AP femur
  * Lauenstein Lateral
  * Cross-Table Lateral (only at the first visit at 5-7 years)
  As a single composite radiographic outcome, the percent of subjects with radiolucencies greater than 2 mm in any zone, acetabular cup migration greater than 4 mm, change in cup inclination greater than 4 degrees or osteolysis at the time of last radiographic assessment will be reported.
Adverse Events | First visit at 5-7 years (1825- 2919 days); Minimum 8-years (2920-3649 days); Minimum 10-years (3650-4015days)
  Subjects who consent to participate in this trial have already had their index surgery for implantation of the study hip; however, potential adverse events may still occur and will be captured at each follow-up visit.
Device survivorship | 5-years, 6-years, 7-years, 8-years, and 9-years
  Device survivorship will be estimated with a Kaplan-Meier survivorship analysis at years 5 through 9 post-operatively

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sacramento, California
  - Denver, Colorado
  - Winston-Salem, North Carolina
  - Orthopedic One, Columbus, Ohio
  - Alexandria, Virginia